CLINICAL TRIAL: NCT03759314
Title: Identification of Risk Patients in Emergency Medical Services
Status: Completed | Type: Observational
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: University of Helsinki (Other)
Responsible Party: Principal Investigator, Marja Mäkinen, Researcher, Helsinki University Central Hospital
Other Study IDs: §50, 27.3.2018
Record Dates: First submitted 2018-11-15; First posted 2018-11-29 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2022-01

CONDITIONS: Malnutrition; Falling; Cognitive Impairment
Keywords: EMS; elderly; nutrition; falling; cognitive functioning
MeSH Terms: conditions — Malnutrition; Cognitive Dysfunction | interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observation — to use a simple screening tool to find out the risk of falling, the nutritional status and the level of cognitive functioning activity

SUMMARY:
Background: Inadequate nutrition has been associated with growing risk of falling and impaired ability in elderly patients. Falling is a significant threat to the health of the elderly. It is estimated that one third of people over the age of 65 experience at least one falling each year. Over 60% of the falls cause serious injury or disability. Adequate nutrition increases the muscle strength of the elderly. Therefore, determining and managing the nutrition level is important for preventing falling. As far as we know emergency medical services has never before reported being a part of prevention by performing risk identification.

DETAILED DESCRIPTION:
Aim: The purpose of the study is to assess whether it is possible to use a simple screening tool to find out the risk of falling, the nutritional status and the level of cognitive functioning activity when the EMS faces the elderly over the age of 70 years. In addition, the flow of information between primary care and emergency services and nutritionists is examined.

Material and method: Identification of poor nutrition is carried out in the Helsinki University hospital area. All people over the age of 70 requiring ambulance transport will be included in the study for 4 months during 2018. A structured electronic form is used to identify the malnutrition, the level of cognitive functioning activity and the risk of falling. The assessment is performed during the transport. The data is analyzed by the SPSS statistical program both by descriptive and statistical significance by looking at the methods suitable for the data.

Conclusion: The information produced by the research aims to develop (a) Identifying in the ambulance those patients who are at risk; and (b) activating nursing staff and nutritionists and, by means of these measures, increase the number of patients receiving effective nutrition therapy.

ELIGIBILITY:
Inclusion Criteria:

* All people over the age of 70 requiring ambulance transport will be included in the study for 4 months during 2018.

Exclusion Criteria:

-

Ages: 70 Years to 104 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All people over the age of 70 requiring ambulance transport will be included in the study for 4 months during 2018 in the Helsinki University hospital area.
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2022-01-28 (Actual); Study Completion 2022-01-28 (Actual)

PRIMARY OUTCOMES:
Identifying in the ambulance those patients who are at risk (over 3 points in a single section) | Through study completion an average of 12 months
  to use a simple screening tool to find out the risk of falling, the nutritional status and the level of cognitive functioning activity when the EMS faces the elderly over the age of 70 The risk-screening tool is based on valid scales. RISK SCREENING TOOL;
  Risk of falling:
  Prediction of falls (4 items, 0-3 points) Self-reporting of falls over a 12-month period (3 items, 0-3 points)
  Malnutrition Risk:
  Home care and meal services (Yes, No) Nutritional status (4 items, 0-3 points) Effect of the diseases on nutrition (4 items, 0-3 points) Age (1 item, 1 point)
  Delirium and cognitive functioning:
  Alertness / memory / attention deficit / symptoms (4 items, 0-3 points)
  Complete when:
  > 70 years patient The patient's physical state allows. Mostly completed during transport (no need to add actual time on scene). Possible risk points are reported at donation to the emergency department.

OTHER OUTCOMES:
Identifying in the ambulance those patients who are at risk (total scores over sections) | Through study completion an average of 12 months
  Subscales are combined to compute a total score, if more than three points in total, the patient is considered to be a risk patient.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Emergency Medicine and Services, Helsinki University Hospital and Helsinki University, Helsinki, Finland, Helsinki, Helsinki Usimaa, Finland

IPD SHARING:
Plan to Share IPD: Undecided